CLINICAL TRIAL: NCT06358131
Title: Propofol Versus Midazolam in Sedation for Upper and Lower Gastrointestinal Endoscopy.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Gameel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R.21.10.1493
Record Dates: First submitted 2023-05-26; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-05

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol arm (Active Comparator)
  Interventions: Device: Endoscopy
- midazolam arm (Active Comparator)
  Interventions: Device: Endoscopy

INTERVENTIONS:
Device: Endoscopy — upper and lower endoscopy

SUMMARY:
There has been rapid growth in the number and complexity of gastrointestinal (GI) endoscopic procedures performed during the last decade. To ensure safe and effective upper GI endoscopy, the choice of an appropriate sedative agent is crucial. Sedation usually categorized into four stages: minimal, moderate, deep and general anesthesia. The upper gastrointestinal [GI] endoscopy usually performed under moderate sedation Sedation usually categorized into four stages: minimal, moderate, deep and general anesthesia. The upper gastrointestinal [GI] endoscopy usually performed under moderate sedation. Benzodiazepines still the most common sedative agents used for conscious sedation, either solely or in combination with opioids for upper GI endoscopy. Propofol is a hypnotic drug used for induction of anesthesia with short half-life that permits rapid patient recovery and discharge. Thus, its use is for upper GI endoscopy was adopted in many endoscopy centers. So we are going to Evaluate all adverse events related to anesthesia; in patients recruited for upper and lower endoscopy and compare between propofol and midazolam based anesthesia associated adverse events.Also we are going to Evaluate patient and endoscopist satisfaction as regarding propofol and midazolam anesthesia.

ELIGIBILITY:
Inclusion Criteria:

Age18 to 80 American Society of Anesthesiologists (ASA) class I-II Informed consent. Patients scheduled for upper and lower endoscopy.

Exclusion Criteria:

Chronic use of drugs as benzodiazpines, neuroleptics and anticonvulsants for more than 30 days.

Hypersensitivity reactions to drugs used in the study. Psychiatric patients. Pregnancy. Being submitted to endoscopy as an emergency procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate all adverse events related to anesthesia; in patients recruited for upper and lower endoscopy and compare between propofol and midazolam based anesthesia associated adverse events. | 2 years

SECONDARY OUTCOMES:
Evaluate patient and endoscopist satisfaction as regarding propofol and midazolam anesthesia. | 2 years
  visual analog scale

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura University, Al Mansurah, Dakhlia
  - MansouraU, Al Mansurah